CLINICAL TRIAL: NCT04362293
Title: Reduced Intensity Related Donor Peripheral Blood Derived Hematopoietic Progenitor Cell Transplantation for Patients With Severe Sickle Cell Disease
Brief Title: Reduced Intensity Transplantation for Severe Sickle Cell Disease
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: We are holding enrollment, due to some recent SAEs.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCDHCT
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea; Azathioprine; Alemtuzumab; Whole-Body Irradiation; Sirolimus; Thiotepa; plerixafor; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Matched Sibling Donor (MSD) (Experimental): Patients with a suitable HLA matched sibling donor (MSD) will be enrolled on the MSD arm.
  Interventions: Drug: hydroxyurea, azathioprine, alemtuzumab, thioptepa, low dose total body irradiation and sirolimus
- Haploidentical (HAPLO) (Experimental): Patients without an eligible MSD who have a suitable haploidentical (HAPLO) donor available will be enrolled on the HAPLO arm of the study.
  Interventions: Drug: hydroxyurea, azathioprine, alemtuzumab, thiotepa, plerixafor, low dose total body irradiation, cyclophosphamide and sirolimus

INTERVENTIONS:
Drug: hydroxyurea, azathioprine, alemtuzumab, thioptepa, low dose total body irradiation and sirolimus — The conditioning regimen will consist of hydroxyurea (30mg/Kg) and azathioprine (3mg/Kg) by mouth daily from day -60 to day -8, alemtuzumab subcutaneously daily for 5 days (0.03mg/kg on Day -7, 0.1mg/kg on Day -6, 0.3mg/kg on days -5 to -3), thiotepa intravenously (10mg/Kg) on day -3 and low dose total body irradiation (TBI) 200 cGY on day -2 with gonadal shielding (if possible). The HSCT graft will be G-CSF mobilized PBSCs with minimum CD34+ of 5 x10^6/kg recipient weight.
  GVHD prophylaxis will be sirolimus with a loading dose 3 mg/m2 on day -1. Sirolimus dose will be adjusted to maintain a target trough level 5-15 ng/mL. Low dose donor lymphocyte infusions will begin on day +28 and continue till donor lymphocyte chimerism reaches at least 90% donor.
  Arms: Matched Sibling Donor (MSD)
Drug: hydroxyurea, azathioprine, alemtuzumab, thiotepa, plerixafor, low dose total body irradiation, cyclophosphamide and sirolimus — The conditioning regimen will consist of hydroxyurea (30mg/Kg) and azathioprine (3mg/Kg) by mouth daily from day -60 to day -8, alemtuzumab subcutaneously daily for 5 days (0.03mg/kg on Day -7, 0.1mg/kg on Day -6, 0.3mg/kg on days -5 to -3), thiotepa intravenously (10mg/Kg) on day -3, plerixafor (0.24mg/Kg) subcutaneously every 12 hours on days -3 and -2 and low dose total body irradiation (TBI) 200 cGY on days -2 and -1 with gonadal shielding (if possible). The HSCT graft will be G-CSF mobilized PBSCs with minimum CD34+ of 5 x10^6/kg recipient weight.
  GVHD prophylaxis will be cyclophosphamide (50mg/Kg) intravenously on days +3 and +4 and sirolimus with a loading dose 3 mg/m2 starting on day +5. Sirolimus dose will be adjusted to maintain a target trough level 5-15 ng/mL. Low dose donor lymphocyte infusions will begin on day +28 and continue till donor lymphocyte chimerism reaches at least 90% donor.
  Arms: Haploidentical (HAPLO)

SUMMARY:
This study is being done to test a transplant method that may have fewer side effects (or less toxic, less harmful) than conventional high dose chemotherapy conditioning-based transplants for children and young adults with Sickle Cell Disease (SCD). Patients less than or equal to 25 years old with SCD who would likely benefit from allogeneic hematopoietic cell transplantation (HCT) will be included in this study. Patients with a suitable HLA matched sibling donor (MSD) will be enrolled on the MSD arm while patients without an eligible MSD who have a suitable haploidentical (HAPLO) donor available will be enrolled on the HAPLO arm of the study.

Primary Objective

To assess the donor T-cell chimerism at 1-year post transplant in each respective arm (MSD, HAPLO) of the trial.

Secondary Objectives

* Assess the overall survival and 1-year, 2-year and 3-year post-transplant graft versus host disease (GVHD)-free SCD-free survival.
* Estimate the primary and secondary graft rejection rate at 1-year, 2-year and 3-year post- transplant.
* Estimate the incidence and severity of acute and chronic (GVHD).
* Estimate the incidence of SCD recurrence after transplant
* Assess the neutrophil and platelet recovery kinetics post-transplant.

Exploratory Objectives

* Record immune reconstitution parameters, including chimerism analysis, quantitative lymphocyte subsets, T cell receptor excision circle (TREC) analysis, V-beta spectratyping, and lymphocyte phenotype and function.
* Conduct longitudinal examination of impact of HCT on patient health-related quality of life (HRQL) and adjustment, and parental adjustment.
* Examine impact of HCT on patient cognitive and academic function.
* Determine factors that influenced the decision to undergo HCT, explore perceptions of the HCT experience, and assess decisional satisfaction/regret.
* Develop and evaluate an objective/quantitative imaging biomarker to assess organ (liver and heart) function/disease status and changes following HCT.
* Develop and evaluate an objective/quantitative imaging biomarker to determine cerebral blood flow and oxygen extraction fraction following HCT.

DETAILED DESCRIPTION:
This is a prospective single center phase II study of a reduced intensity conditioning based hematopoietic cell transplant for patients with sickle cell disease. In this study, patients with SCD who would be expected to benefit from an allogeneic HCT will receive an unmanipulated peripheral blood derived hematopoietic stem and progenitor cell (HSPC) graft from either an MSD or HAPLO donor after a reduced intensity conditioning regimen comprising of alemtuzumab, thiotepa and low dose total body irradiation. All patients will receive a pre-conditioning phase comprising of hydroxyurea and azathioprine to reduce the risk of graft rejection. GVHD prophylaxis will consist of sirolimus. Patients on the HAPLO arm will also receive two doses of post-transplant cyclophosphamide. All patients will receive regularly scheduled low dose donor lymphocyte infusions till donor lymphocyte chimerism reaches at least 90% donor. The main objective of this study is to improve graft function and immune reconstitution after a reduced intensity conditioning based transplant.

ELIGIBILITY:
Inclusion Criteria for Transplant Recipient

* Age less than or equal to 25 years.
* Patients with a suitable HLA-matched sibling donor (MSD) can be enrolled on MSD arm of the trial. Patients with single haplotype matched (≥ 3 of 6) family member donor can be enrolled on HAPLO arm of the trial, if they do not have a suitable HLA-matched sibling donor (MSD) available for progenitor cell donation.
* Patients with SCD (any genotype) who meet any ONE of the following criteria:

  1. History of an abnormal transcranial Doppler measurement defined as TCD velocity ≥ 200 cm/sec by the non-imaging technique (or ≥ 185 cm/sec by the imaging technique) measured at a minimum of two separate occasions.
  2. History of cerebral infarction on brain MRI (overt stroke, or silent stroke if ≥3 mm in one dimension, visible in two planes on fluid-attenuated inversion recovery T2- weighted images).
  3. History of two or more episodes of acute chest syndrome (ACS) in the 2-years period preceding enrollment.
  4. History of two or more SCD pain events requiring treatment with an opiate or IV pain medication (inpatient or outpatient) in the last 12 months.
  5. History of any hospitalization for SCD pain or ACS while receiving hydroxyurea treatment in the last 12 months.
  6. History of two or more episodes of priapism (erection lasting ≥4 hours or requiring emergent medical care).
  7. Administration of regular RBC transfusions (≥8 transfusions in the previous 12 months).
  8. At least two episodes of splenic sequestration requiring red blood cell transfusion or splenectomy after at least one episode of splenic sequestration.

Exclusion Criteria for Transplant Recipient

* Karnofsky or Lansky performance score <60.
* Pregnant or breastfeeding patients.
* Uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms) within 1 month prior to conditioning. Patients with febrile illness or suspected minor infection should await clinical resolution prior to starting conditioning. Patients with confirmed seropositivity or positive NAAT for HIV are excluded.
* Serum conjugated (direct) bilirubin >3x upper limit of normal for age as per local laboratory. Participants with hyperbilirubinemia or elevated AST as the result of hyperhemolysis, or a severe drop in hemoglobin post blood transfusion, are not excluded as long as it downtrends and return to acceptable limits subsequently.
* Left ventricular shortening fraction <25% or ejection fraction <40% by echocardiogram.
* Estimated creatinine clearance less than 50 mL/min/1.73m2.
* Diffusion capacity of carbon monoxide (DLCO) <35% (adjusted for hemoglobin). Baseline oxygen saturation <85% or PaO2 <70.
* Presence of anti-donor specific HLA antibodies unresponsive to desensitization as defined below.

HLA antibody presence and specificity will be determined by solid phase immunoassays. An anti-donor specific HLA antibody test will be considered positive when the mean fluorescence intensity (MFI) is:

* >1,000 for donor specific antibodies to HLA-A, -B, and DRB1. or
* >2,000 for donor specific antibodies to HLA-C, DQB1 and DPB1.

A participant with presence of anti-donor specific HLA antibodies may be provisionally enrolled on the study if desensitization (see Appendix H) is begun concurrently with pre-conditioning. Response to desensitization will be defined as:

* decreasing anti-donor specific HLA antibody titer with an MFI of less than 5,000 and
* negative C1q-binding anti-HLA antibody assay.

Inclusion Criteria for Donor

* An HLA-matched sibling donor for MSD arm and at least single haplotype matched (≥ 3 of 6) family member for HAPLO arm.
* HIV negative.
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* Not breast feeding.
* Donor should not have clinically significant hemoglobinopathy. Donors with sickle cell trait are acceptable.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Donor T-cell chimerism at 1-year post transplant in each respective arm (MSD, HAPLO) of the trial. | 1 year after HCT
  Number of participants who have achieved donor T-cell chimerism greater than 60% by 1-year post transplant will be reported. The rate of success will be checked for in each arm after the first 10 evaluable patients have been enrolled and followed for up to 1 year.

SECONDARY OUTCOMES:
Overall survival and 1-year, 2-year and 3-year post-transplant graft versus host disease (GVHD)-free SCD-free survival. | Up to 3 years after HCT
  Graft versus host disease (GVHD)-free SCD-free survival in each arm of the trial will be calculated at 1-year, 2-year and 3-year post-transplant and reported as a percentage of the enrolled patients.
Graft rejection rate. | Up to 3 years after HCT
  Primary and secondary graft rejection rate at 1-year, 2-year and 3-year post- transplant in each arm or the trial will be calculated and reported as a percentage of the enrolled patients.
Incidence and severity of acute and chronic (GVHD). | Up to 3 years after HCT
  The incidence and severity of acute and chronic (GVHD) in each arm or the trial will be calculated and reported as a percentage of the enrolled patients.
Incidence of SCD recurrence after transplant. | Up to 3 years after HCT
  The incidence of SCD recurrence after transplant in each arm or the trial will be calculated and reported as a percentage of the enrolled patients.
Neutrophil and platelet recovery. | Up to 6 months after HCT
  Number of patients who engraft their neutrophils and platelets by 6 months in each arm or the trial will be calculated and reported as a percentage of the enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Sharma, MBBS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- [Derived] Sharma A, Selukar S, Bi Y, Merlocco A, Morin CE, Goode C, Rai P, Towbin JA, Hankins JS, Gottschalk S, Triplett B, Johnson JN. Impact of hematopoietic cell transplantation on myocardial fibrosis in young patients with sickle cell disease. Blood. 2024 Aug 8;144(6):672-675. doi: 10.1182/blood.2023023028. PMID 38691679
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols